CLINICAL TRIAL: NCT02498041
Title: Study to Compare the Efficacy and Patient Tolerance of Ultrathin Nasal Endoscopy to Detect Barrett's Esophagus Compared With Conventional Endoscopy to Inform a Future Multicentre Screening Trial
Brief Title: The Efficacy and Patient Tolerance of Ultrathin Nasal Endoscopy to Detect Barrett's Oesophagus
Acronym: NOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Senior Clinician Scientist and Consultant Gastroenterologist, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UCambridge
Record Dates: First submitted 2015-07-07; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Barrett's Esophagus; Dyspepsia
Keywords: Ultrathin Nasal Endoscopy; Barrett's Esophagus; Transnasal Endoscopy
MeSH Terms: conditions — Barrett Esophagus; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transnasal Endoscopy (Experimental): Unsedated transnasal endoscopy with biopsies
  Interventions: Procedure: Transnasal Endoscopy; Device: Office-based disposable transnasal endoscopy Endosheath; Procedure: Esophageal biopsies
- Standard Gastroscopy (Active Comparator): Standard endoscopy with biopsies. Patients will decide whether they prefer to have endoscopy with intrevenous sedation or with local anaesthetic only
  Interventions: Device: Standard upper GI endoscopy; Procedure: Esophageal biopsies

INTERVENTIONS:
Procedure: Transnasal Endoscopy — Experimental procedure with transnasal endoscopy for the first 80% of the patients (n=90). The examination is limited to the esophagus and the proximal stomach.
  Other Names: EG530N; Fujinon, Fujifilm, Valhalla, NY
  Arms: Transnasal Endoscopy
Device: Office-based disposable transnasal endoscopy Endosheath — Experimental procedure with portable, disposable transnasal endoscopy for the last 20% of patients only (n=25). The examination is limited to the esophagus and the proximal stomach.
  Other Names: Endosheath; Vision® Sciences, Inc, New York, USA
  Arms: Transnasal Endoscopy
Device: Standard upper GI endoscopy — Upper GI endoscopy with standard gastroscope.
  Other Names: Esophago-gastro-duodenoscopy
  Arms: Standard Gastroscopy
Procedure: Esophageal biopsies — 2 research biopsies taken if endoscopic evidence of columnar-lined esophagus
  Other Names: Research biopsies

SUMMARY:
This study evaluates the diagnostic accuracy, safety and acceptability of transnasal endoscopy (TNE) for a diagnosis of Barrett's esophagus (BE). This is a cross-over randomised trial, whereby patients receive two endoscopic procedures 2-4 weeks apart and will be randomised to receive either TNE or standard endoscopy followed by the other procedure.

DETAILED DESCRIPTION:
Background: The incidence of esophageal adenocarcinoma (EAC) has drammatically increased in the Western World in the last 30 years. Furthermore it often presents in the late stages and the prognosis remains poor with an overall 5-year survival of 10-15%. Early detection is possible since most cases of EAC develop from a precursor condition, Barrett's esophagus (BE), via a metaplasia-dysplasia-adenocarcinoma sequence. BE can be diagnosed with an upper GI endoscopy.

Un-sedated trans-nasal endoscopy (TNE) may be safer and less expensive than standard endoscopy (SE) for detecting BE. Emerging technologies require robust evaluation before routine use.

Objective: To evaluate the sensitivity, specificity, and acceptability of TNE in diagnosing BE compared with those of SE.

Design:Prospective, randomized, crossover study

Setting:Single, tertiary-care referral center.

Patients: patients with BE or those referred for diagnostic assessment will be enrolled consecutively .

Intervention: All patients will undergo TNE followed by SE or the reverse. Spielberger State-Trait Anxiety Inventory, short-form questionnaires, a visual analogue scale, and a single question addressing preference for endoscopy type will be administered.

Main Outcome Measurements: Diagnostic accuracy for BE and tolerability of TNE and SE.

The primary aim of this study is to evaluate the sensitivity and specificity of ultrathin endoscopy in diagnosing BE (using standardised endoscopic and histopathological criteria) compared with the gold standard white light conventional endoscopy.

The secondary aims include to assess the acceptability, optical quality and safety of the two interventions.

The study will consist of two phases. In a first large phase 80% of the target (90 patients) we will evaluate conventional TNE (Fujinon). In a second phase the remaining of the patients (25) will be evaluated with a disposable office-based system (Endosheath).

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 18 years and <75 years
2. Patients who have given informed consent and who are capable of filling in the questionnaire.
3. Patients requiring endoscopy for dyspepsia or follow-up evaluation and patients with a prior diagnosis of BE (defined as minimum Barrett's length of 2cm - according to M level of Prague C & M classification) with specialized intestinal metaplasia on histological confirmation.

Exclusion Criteria:

1. Previous upper GI tract or upper respiratory tract surgery or known upper GI tract abnormality (e.g. pharyngeal pouch).
2. Coagulopathy or on anticoagulants
3. Active or severe cardiopulmonary disease or liver disease
4. Active GI bleeding
5. Patients with alarm symptoms referred to the fast track service and any patient with dysphagia
6. Patients requiring possible endoscopic therapy
7. Patients with high-grade dysplasia or intramucosal carcinoma in BE requiring extensive evaluation and biopsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Endoscopic Diagnostic Accuracy for Barrett's esophagus | 2 weeks
  Sensitivity and specificity for detecting BE using ultrathin endoscopy when compared to gold standard conventional endoscopy will be calculated along with 95% Pearson-Clopper confidence intervals.

SECONDARY OUTCOMES:
Optical accuracy | 2 weeks
  Interobserver agreement for an endoscopic diagnosis of BE by different endoscopic interventions. The optical quality of ultrathin endoscopy will be compared with conventional endoscope by using a 10-cm VAS, where 10 is excellent and 0 is poor.
Histological diagnosis of Barrett's esophagus | 2 weeks
  Yield of intestinal metaplasia in the biopsies taken at both procedures. The presence of intestinal metaplasia in research biopsies taken using ultrathin endoscopy will be compared with standard endoscopy.
Patient acceptability | 12 weeks
  The overall acceptability for each procedure will be measured by State-Trait Anxiety inventory, Visual Analogue Scale and SF6 and the choice of procedure in future.
Adverse events | 1 week
  Any adverse events reported by the patient in the week following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Fitzgerald, MD, Principal Investigator — University of Cambridge; M. Kareem Shariff, MRCP, Principal Investigator — University of Cambridge; Massimiliano di Pietro, MD, Principal Investigator — University of Cambridge